CLINICAL TRIAL: NCT00134823
Title: Improving Pediatric Safety and Quality With Health Care IT
Brief Title: Improving Pediatric Safety and Quality With Health Care Information Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Timothy G Ferris, Mass General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2004-P-002027; HS015002-01 (Other Grant/Funding Number: AHRQ)
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Medication Errors; Medical Records Systems, Computerized; Patient Safety; Quality Improvement
Keywords: Parent Experience of Care; Quality Improvement; Medication Errors; Abnormal Lab Values; Guideline Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dosing decision support (Experimental): weight based dosing decision support
  Interventions: Other: weight based dosing decision support
- no decision support (No Intervention): no weight based dosing decision support

INTERVENTIONS:
Other: weight based dosing decision support — weight based dosing decision support
  Arms: dosing decision support

SUMMARY:
This study includes four projects aimed to improve the quality and safety of pediatric care through the implementation of four clinical decision support services in the electronic health record (EHR). The four projects will measure the effect of each clinical decision support feature including: weight-based dosing; smart forms for chronic conditions; guideline reminders; and a results manager to track abnormal lab result follow-up.

Hypothesis: Implementation of the clinical decision support features will decrease medication errors and adverse drug events, assist physicians in adhering to clinical practice guidelines and protocols for certain chronic illnesses, improve physician follow-up for abnormal lab results, and overall improve the safety and quality of pediatric clinical practice.

DETAILED DESCRIPTION:
please see description above

ELIGIBILITY:
Inclusion Criteria:

* Partners-affiliated pediatric practice providers utilizing Longitudinal Medical Record (LMR), which is an electronic health record system. Also the parents of the patients of the above noted pediatric providers.

Exclusion Criteria:

* Non-Partners providers, or Partners providers who do not use LMR. Parents of patients not seen by Partners-affiliated pediatric providers who use LMR.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5420 (Actual)
Dates: Start 2005-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Impact on rates of medication errors | 1 year
  difference in weight related medication prescribing errors by drug class

CONTACTS AND LOCATIONS:
Overall Officials: Timothy G Ferris, MD, MPH, Principal Investigator — Massachusetts General Hospital, Partners Healthcare System Inc.
Locations (1):
- Massachusetts General Hospital/Partners HealthCare, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bourgeois FC, Linder J, Johnson SA, Co JP, Fiskio J, Ferris TG. Impact of a computerized template on antibiotic prescribing for acute respiratory infections in children and adolescents. Clin Pediatr (Phila). 2010 Oct;49(10):976-83. doi: 10.1177/0009922810373649. Epub 2010 Aug 19. PMID 20724348
- [Derived] Co JP, Johnson SA, Poon EG, Fiskio J, Rao SR, Van Cleave J, Perrin JM, Ferris TG. Electronic health record decision support and quality of care for children with ADHD. Pediatrics. 2010 Aug;126(2):239-46. doi: 10.1542/peds.2009-0710. Epub 2010 Jul 19. PMID 20643719